CLINICAL TRIAL: NCT06076057
Title: Vital Signs Monitoring of Emergency Responders in Different States
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2021CXGC011301
Record Dates: First submitted 2023-09-13; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Heart Rate Monitoring
Keywords: Vital Signs; Respiration; transcutaneous oxygenation; end-expiratory carbon dioxide
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- 8:00 Measurement team: At 08:00 , monitoring respiratory rate, pulse rate, oxygen saturation, body position, thoracic and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration, partial pressure of transcutaneous oxygen, and partial pressure of transcutaneous carbon dioxide.
  Interventions: Diagnostic Test: vital signs monitoring
- 10:30 Measurement team: At 10:30 , monitoring respiratory rate, pulse rate, oxygen saturation, body position, thoracic and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration, partial pressure of transcutaneous oxygen, and partial pressure of transcutaneous carbon dioxide.
  Interventions: Diagnostic Test: vital signs monitoring
- 16:30 Measurement team: At 16:30 , monitoring respiratory rate, pulse rate, oxygen saturation, body position, thoracic and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration, partial pressure of transcutaneous oxygen, and partial pressure of transcutaneous carbon dioxide.
  Interventions: Diagnostic Test: vital signs monitoring
- high altitude environment: In high altitude environments, monitoringRespiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration
  Interventions: Diagnostic Test: vital signs monitoring
- limited space: In limited space environments, monitoringRespiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration
  Interventions: Diagnostic Test: vital signs monitoring
- electrified operation: In electrified operation , monitoringRespiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration
  Interventions: Diagnostic Test: vital signs monitoring
- work site: In work site , monitoringRespiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration
  Interventions: Diagnostic Test: vital signs monitoring

INTERVENTIONS:
Diagnostic Test: vital signs monitoring — Monitoring of vital signs using portable respiratory sleep monitors, NoxT3, carbon dioxide monitors, transcutaneous oxygen and carbon dioxide partial pressure monitors

SUMMARY:
The goal of this observational study is to learn about emergency responder in different states. The main questions it aims to answer are:

* Ten vital signs and behavioral parameters in different states (quiet, after post, after physical training) including: respiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration, partial pressure of transcutaneous oxygen, and partial pressure of transcutaneous carbon dioxide.
* Eight vital signs and behavioral parameters in different environments (altitude, confined space, energized work, job site) including: respiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), and partial pressure of end-expiratory CO2 concentration.

Participants will normal operating conditions, the researcher collects vital sign information.

DETAILED DESCRIPTION:
1. General information: name, age, height, weight, place of origin, smoking history, and whether or not they snore.
2. 10 vital signs and behavioral parameters in different states (quiet, after duty, after physical training), including: respiratory rate, pulse rate, oxygen saturation, body position, chest and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), partial pressure of end-expiratory CO2 concentration, partial pressure of transcutaneous oxygen, partial pressure of transcutaneous carbon dioxide.
3. 8 vital signs and behavioral parameters in different environments (overhead, confined space, energized work, work site), including: respiratory rate, pulse rate, oxygen saturation, body position, thoracic and abdominal respiratory movements, electromyography (EMG), electroencephalogram (EEG), and partial pressure of end-expiratory CO2 concentration.

ELIGIBILITY:
Inclusion Criteria:

* No history of coronary heart disease, hypertension, asthma, upper respiratory tract infection, decompression sickness, or anemia.

Voluntarily participated in this study and signed an informed consent form

Exclusion Criteria:

* Patients with severe heart disease and arrhythmia; patients with vital organ failure; patients with significant generalized edema; patients with dermatologic disease and generalized skin breakdown; and patients with vascular disorders of the limbs.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Frontline National Grid Emergency Responders
Sampling Method: Non-Probability Sample
Enrollment: 135 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
respiratory rate | 3 month
  Breaths per minute
heart rate | 3 month
  beats per minute
blood oxygen saturation | 3 month
  Concentration of oxygen in the blood
electromyography | 3 month
  Measurement and analysis of electromyographic signals emitted during muscle contraction
electroencephalogram | 3 month
  Collecting brainwave signals，Analyze the EEG for abnormalities
Partial pressure of end-expiratory CO2 concentration | 3 month
  Measurement of the partial pressure of CO2 in exhaled gas at the end of expiration
transcutaneous partial pressure of oxygen | 3 month
  Measurement of the partial pressure of oxygen at the skin surface, thus indirectly reflecting the state of tissue oxygenation
Percutaneous carbon dioxide partial pressure | 3 month
  Indirectly reflecting the partial pressure of carbon dioxide by measuring the pH of the skin surface

CONTACTS AND LOCATIONS:
Overall Officials: luan xiaorong, Study Chair — Shandong University Qilu Hospital
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No